CLINICAL TRIAL: NCT01304108
Title: Spreading and Improving DVT Prophylaxis at Mayo Clinic (DVT-P-Spread)
Brief Title: Improving Venous Thromboembolism Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Timothy Morgenthaler, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-006359
Record Dates: First submitted 2010-07-09; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Venous Thromboembolism; Delivery of Health Care; Quality Improvement
Keywords: Venous Thromboembolism; Delivery of Health Care; Quality Improvement; Evidence-Based Practice
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Order Set (Experimental): Insertion of VTE-P Order Set "tollgate" in all active admission and transfer orders.
  Interventions: Other: VTE-P Tollgate
- Clinical Decision Support Pop-up (Experimental): Deploy rules-based pop-up that reminds ordering clinicians when patients do not have an active VTE-P plan.
  Interventions: Other: BLAZE Pop up
- Usual Care (Active Comparator): Usual care, without the experimental additions
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: VTE-P Tollgate — Add VTE-P tollgate order set that requires a decision regarding VTE-P for every patient admitted or transferred in our hospital system
  Arms: Order Set
Other: BLAZE Pop up — Develop and deploy a rules-based popup that reminds prescribers interfacing with the orders system when a patient does not have an active VTE-P plan.
  Arms: Clinical Decision Support Pop-up
Other: Usual Care — No addition to the baseline system for care
  Arms: Usual Care

SUMMARY:
Preventing the formation of blood clots in the veins so they do not injure leg veins or travel to the lungs, also called venous thromboembolism prophylaxis (VTE-P) is an essential component of safe in-patient care, yet it is deployed sub-optimally in many hospitals, including The investigators own. Two prior VTE-P improvement projects were completed at Mayo Clinic hospitals, one in the Department of Medicine, and the other in selected divisions of the Department of Surgery. Both projects resulted in marked improvement in the percentage of patients receiving appropriate VTE-P. This project seeks to utilize the lessons learned from these two pilots along with known best practices for "spreading" to deploy methods that enhance VTE-P to the entire hospitalized population. The investigators seek appropriate VTE-P rates exceeding 95%.

DETAILED DESCRIPTION:
Venous thromboembolism prophylaxis (VTE-P) is an essential component of safe in-patient care, yet it is deployed sub-optimally in many hospitals, including our own. Two prior VTE-P improvement projects were completed at Mayo Clinic hospitals, one in the Department of Medicine, and the other in selected divisions of the Department of Surgery. Both projects resulted in marked improvement in the percentage of patients receiving appropriate VTE-P. This project seeks to utilize the lessons learned from these two pilots along with known best practices for "spreading" to deploy methods that enhance VTE-P to the entire hospitalized population. The investigators seek appropriate VTE-P rates exceeding 95%. This began as a quality improvement project. The investigators have taken baseline measures of VTE-P rates in our hospitals, intervened with various electronic prompts to use appropriate VTE-P, and have and will re-measure VTE-P rates. The investigators intend to present and publish our methods and results so that lessons learned may be shared and applied elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with age > 17 years old

Exclusion Criteria:

* Outpatients
* Inpatients with age less than or equal to 17 years old

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
% of in patients with an appropriate VTE prophylaxis plan | Baseline to 1 month
  The investigators will measure the number of patients in a statistically valid random sample of hospitalized patients who have a VTE-prophylaxis plan consistent with current recommendations.

SECONDARY OUTCOMES:
Clinically significant complications of VTE-P anticoagulant therapy | baseline to 1 month
  The investigators will determine the rate of bleeding complications in inpatients using a statistically valid random sample of hospitalized patients. The investigators will also determine the rate of procedure delays due to VTE-P related anticoagulation.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgenthaler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States